CLINICAL TRIAL: NCT01809548
Title: Early Introduction of Solid Foods in Preterm Infants: Effects on Growth, Atopy and Neurodevelopment
Brief Title: Preterm Infants on Early Solid Foods
Acronym: PIES-Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, Assoc.Prof.PD. MD, MSc, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIES001
Record Dates: First submitted 2013-03-01; First posted 2013-03-12 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Infant, Very Low Birth Weight; Growth Failure
Keywords: complementary feeding; premature infant; body composition; atopy; neurodevelopmental outcome; obesity
MeSH Terms: conditions — Failure to Thrive; Premature Birth; Obesity

STUDY DESIGN:
Masking Description: After interim analysis switch from prospective randomised to baseline adaptive randomised controlled - stratified according birthweight below /equal 800g and equal/more than 801 grams.
  After an interim analysis 1/2019: During the whole study period we had a very low drop out rate of 11% so far. Therefore we adapt the sample size calculation from the anticipated 30% drop out rate to an one-to-one replacement for dropouts + a surplus of 5 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early complementary feeding group (Experimental): Early intervention group:
  Introduction of early complementary feedings between the 10th -12th week of gestation corrected for prematurity
  Interventions: Other: Early intervention group
- Late complementary feeding group: (Experimental): Late intervention group:
  Introduction of late complementary feedings between the 16th and 18th week of life corrected for prematurity
  Interventions: Other: Late intervention group

INTERVENTIONS:
Other: Early intervention group — solid food will be introduced between week 10 and 12
  Other Names: commercially available solid food
  Arms: Early complementary feeding group
Other: Late intervention group — solid food is introduced between 16-18th week of gestation corrected for prematurity
  Other Names: commercially available solid food
  Arms: Late complementary feeding group:

SUMMARY:
Introduction: Preterm infants with a birth weight less than 1500 grams have special nutritional needs in comparison to full-term neonates. During their stay in the neonatal intensive care unit an increased supply with energy, protein and electrolytes is necessary to establish adequate growth. After discharge from the hospital special breast milk supplements or post discharge formulas are available to cover the special nutrient requirements. Complementary feeding in preterm infants is an unexplored field so far and nutritional concepts for the first year of life are not available. Data concerning the optimal time for starting solid foods are missing as well as information concerning the ideal composition of complementary food. In this context it is essential to meet the special nutritional needs of "Ex-Preemies" on the one hand and avoid overfeeding and later obesity on the other hand. So far it remains unclear, what the "safe" time point for introduction of solid food to premature infants is and whether this time point influences growth, body composition, neurodevelopmental outcome or the incidence of atopic disease.

DETAILED DESCRIPTION:
Aim: In a prospective, randomized, two arm intervention study- the PIES project- we aim to investigate the impact of different time points of introduction of complementary food on growth, body composition, atopic disease and neurodevelopmental outcome in preterm infant with a birth weight <1500 grams. Furthermore, we want to investigate whether a certain standardized feeding protocol meets the nutritional needs of premature infants, and obtain data on safety and efficacy in this context. Methods: At term infants are stratified according to breastfed or formula fed and randomized in one of the following groups: an EARLY complementary feeding group (introduction of complementary food between the 10th and 12th week of life corrected for term, n=76) and LATE complementary feeding group (introduction of complementary food between the 16th and 18th week of life corrected for term, n=76). The infants will be fed with standardized complementary food in addition to formula or breastfeeding until they are one year corrected for prematurity. In an age dependent step up concept, food boxes are delivered to the parents: five types of standardized food boxes with manifold complementary food according to the infants' age and the ability to tolerate small pieces are available for each child during the study. The standardized complementary feeding regimen allows calculating exact intake of nutrients and therefore will provide information concerning primary and secondary outcome. The follow up phase will last until 5 years of age. Within regular visits anthropometric data (height, head circumference, weight, BMI and z-scores ) and body composition via the PeaPod® system will be gathered. Data on atopy will be assessed by clinical scoring system SCORAD (SCORing Atopic Dermatitis) and the laboratory parameters Fx5(Fx5 test uses six food allergens: wheat, egg, cow's milk, soya, peanut and fish) and IgE (immuneglobulineE). Neurodevelopmental outcome will be assessed at the age of one and two years corrected for term by the Bayley Scales and the K-ABC (Kaufman Assessment Battery for Children). The nutritional concept will be monitored concerning short term safety and efficacy (bone metabolism, iron status, protein- and lipid status) as well as regarding long term outcome (diabetes and obesity markers IGF-1 (Insulin-like growth factor-1, adiponectin and leptin).

With the PIES project we intend to close a gap of knowledge in feeding the premature infant during the first year of life and to understand the impact of complementary feeding on growth, atopy, neurodevelopmental outcome and later obesity.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <1500 gram
* Informed consent

Exclusion Criteria:

Diseases affecting stable growth:

* Gastrointestinal diseases: necrotizing enterocolitis, Hirschsprung disease, chronic inflammatory bowel disease
* Bronchopulmonary dysplasia (BPD) defined as oxygen demand above 36 week gestational age
* Congenital heart diseases
* major congenital birth defects
* chromosomal aberrations

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2013-10; Primary Completion 2020-03-30 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Height: | 1 Year
  To investigate whether a height difference of 5% at one year of age, corrected for prematurity, can be achieved between the early and the late intervention group.
  Height will be measured under standardized conditions in centimeter (cm) at defined times during the first year of life until one year of age corrected for prematurity. Measurements will be done before, within and after intervention in order to demonstrate the changes due to all intervention tools.

SECONDARY OUTCOMES:
neurodevelopmental outcome | 5 years
  To achieve an improvement of neurodevelopmental outcome assessed by Bayley scales and the K-ABC
IGF-1 | 5 years
  To evaluate the risk for later obesity
FX5 | 5 years
  To achieve a reduction in risk for atopic diseases
SCORAD | 5 years
  To achieve a reduction in risk for atopic diseases.
Body composition | 5 years
  To achieve an increase of free fat mass (FFM) in body composition measured with the Peapod.
Vitamin D | 1 year
  To achieve a degree of bone mineralization.
Iron status | 1 year
  To achieve the development of anemia
Leptin | 5 years
  To evaluate the risk for later obesity
BMI | 5 years
  to evaluate anthropometric parameters
weight | 5 years
  to evaluate anthropometric parameters
head circumference | 5 years
  to evaluate anthropometric parameters
z-scores | 5 years
  to evaluate anthropometric parameters

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gsoellpointner M, Eibensteiner F, Thanhaeuser M, Ristl R, Jilma B, Berger A, Haiden N. Effects of early introduction of solid foods on nutrient intake in preterm infants during their 1st year of life: a secondary outcome analysis of a prospective, randomized intervention study. Front Nutr. 2023 May 18;10:1124544. doi: 10.3389/fnut.2023.1124544. eCollection 2023. PMID 37275631